CLINICAL TRIAL: NCT06690918
Title: Risk Factors Contributing to Oral Cancer in Patients at Dr. Hasan Sadikin General Hospital Bandung
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: SURG-202411.01
Record Dates: First submitted 2024-11-04; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Oral Cavity Cancer
Keywords: Oral cavity cancer; Risk factors; Smoking; Alcohol; Betel quid chewing
MeSH Terms: conditions — Mouth Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral cavity cancer group: The inclusion criterion was a confirmed diagnosis of oral cavity cancer undergoing surgical intervention. Patients with oral cancer resulting from metastasis from a primary tumor located in another organ were excluded.
- Control group: The control group consisted of individuals attending the hospital for non-cancer-related conditions matched by age and sex to the case group.

SUMMARY:
Analytical research with a cross-sectional approach was carried out on patients diagnosed with oral cavity cancer who visited our outpatient clinic in Bandung between 2023 and 2024. Data were collected and analyzed using the chi-square test to determine the significance of the relationship between smoking, alcohol consumption, oral hygiene, and betel quid chewing and oral cavity cancer.

DETAILED DESCRIPTION:
This study was conducted using a cross-sectional analytical design, allowing the assessment of the association between various risk factors and oral cavity cancer. This study was conducted at the oncology, ENT, and oral surgery outpatient clinics at our hospital from January 2023 to December 2024. The inclusion criterion was a confirmed diagnosis of oral cavity cancer undergoing surgical intervention. Patients with oral cancer resulting from metastasis from a primary tumor located in another organ were excluded. The control group consisted of individuals attending the hospital for non-cancer-related conditions matched by age and sex to the case group.

Data were collected through structured interviews using a questionnaire designed to obtain information on subject behavior, including smoking, alcohol consumption, betel quid chewing, and oral hygiene practices. Medical records were reviewed to gather additional clinical information and to confirm the diagnosis of oral cavity cancer.

Data were analyzed using SPSS version 25. Descriptive statistics were used to summarize the demographic and clinical characteristics of the study population. The chi-squared test was used to assess the significance of the association between risk factors and the presence of oral cavity cancer. Statistical significance was set at P < 0.05. The study was approved by the Health Research Ethics Committee (registration number DP.04.03/D.XIV.6.5/191/2024).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of oral cavity cancer undergoing surgical intervention.

Exclusion Criteria:

* Oral cancer resulting from metastasis from a primary tumor located in another organ

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted at the oncology, ENT, and oral surgery outpatient clinics of the hospital from January 2023 to December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Risk factors for oral cavity cancer | 3 months
  Risk factors for oral cavity cancer will be listed

CONTACTS AND LOCATIONS:
Overall Officials: Agung Adhariensya, MD, Study Chair — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Universitas Padjajaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No